CLINICAL TRIAL: NCT06339957
Title: Title of Study: Eating Habits and Symptom Severity in Autoimmune Diseases: a Patient Survey
Brief Title: Rheumatology Diet Study
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00006394
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Diet Habit; Rheumatologic Disease; Autoimmune Diseases; Rheumatoid Arthritis; Psoriatic Arthritis; Ankylosing Spondylitis; Dermatomyositis/polymyositis; Sjogren's Syndrome; Systemic Lupus Erythematous; Scleroderma; Fibromyalgia
MeSH Terms: conditions — Feeding Behavior; Collagen Diseases; Autoimmune Diseases; Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing; Dermatomyositis; Sjogren's Syndrome; Scleroderma, Diffuse; Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to collect information on rheumatology patients' dietary habits, autoimmune disease activity, dietary changes, disease symptom improvements, and perceptions on their dietary habits and how it affects their autoimmune disease. The main objective is to see if rheumatology patients change their dietary habits after their diagnosis of an autoimmune disease and if it subjectively improved their disease symptoms. It will also look at rheumatology patients' expectations for their rheumatologist when it comes to dietary advice and what resources they used to choose their new dietary habits. The study also seeks to measure the interest that rheumatology patients have in pursuing dietary changes as a means of controlling the symptoms of their autoimmune disease. It is expected that patients who changed their eating habits to healthier diets such as a Mediterranean diet would report less severe autoimmune disease symptoms. There are limited dietary recommendations for the management of many rheumatological diseases, so this study seeks to assess rheumatology patients' willingness to try dietary modifications, what improvements they had, and why they decide to make these changes in light of limited information.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18 years old) patients
* established UCF Health patients
* diagnosed with rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, dermatomyositis/polymyositis, Sjogren's Syndrome, systemic lupus erythematous, scleroderma, osteoarthritis, or fibromyalgia.

Exclusion Criteria:

* UCF Students, Faculty or Staff
* Children or Young Adults Under the age of 18
* Adults over 65
* Pregnant Women
* Prisoners
* Adults to Unable to Consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants are expected to come from the established rheumatology patient census at the UCF Health Clinics. The research team will identify potential participants via pre-screening the electronic medical records for the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
To determine how diet habits and activity affects autoimmune diseases using the proper statistical tests for the data set such as t-test and ANOVA. | 4 months

SECONDARY OUTCOMES:
To identify if rheumatology patients change their dietary habits after their diagnosis of an autoimmune disease and if it subjectively improved their disease symptoms. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Neha Bhanusali, MD, Principal Investigator — University of Central Florida
Locations (1):
- UCF Health Clinics, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No